CLINICAL TRIAL: NCT03406520
Title: Chlorhexidine-impregnated Sponge Dressing for Prevention of Catheter Exit Site Infection in Incident Peritoneal Dialysis Patients - a Pilot Study
Brief Title: Chlorhexidine Disk for Prevention of Exit-site Infection in Peritoneal Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SRG-NIG#08/2017
Record Dates: First submitted 2018-01-14; First posted 2018-01-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Peritoneal Dialysis Catheter Exit Site Infection
Keywords: peritoneal dialysis; chlorhexidine; exit site infection; tunnel tract infection

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Chlorhexidine-impregnated disk (Experimental): The chlorhexidine-impregnated disk, will be applied to the peritoneal dialysis catheter exit-site and the disk will be changed once a week
  Interventions: Device: Chlorhexidine-impregnated disk

INTERVENTIONS:
Device: Chlorhexidine-impregnated disk — The chlorhexidine-impregnated sponge, named biopatch, is a protective disk (2.5 cm x 0.7 cm), which is hydrophilic polyurethane absorptive foam with chlorhexidine gluconate, in average of 86.8mg per disk
  Other Names: biopatch disk

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of chlorhexidine-impregnated disk in preventing catheter exit-site infection in peritoneal dialysis patients

DETAILED DESCRIPTION:
The primary aim of the study is to examine the exit-site infection rate in patients using chlorhexidine-impregnated dressing.

The participant will be followed up at 2, 6, 12, 24, 36 and 52 weeks of study and during each visit the catheter exit-site will be examined by one of the investigators for any sign of infection or allergic reaction, and questionnaires about satisfaction with use of study material (biopatch) will be asked by a study team member at the 12 week visit of the study. Each participant will be followed up for one year.

ELIGIBILITY:
Inclusion Criteria:

* All adult incident peritoneal dialysis patients between 21 to 90 years old, who are followed up in Singapore General Hospital

Exclusion Criteria:

1. patients who have known history of allergy to chlorhexidine
2. patients who had previous history of peritoneal dialysis catheter exit-site infection
3. patients with mentally challenging conditions who are unable to give the valid consent for the study
4. patients who have been involved in another study for exit site infection

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Exit-site/tunnel infection rate | one year
  Exit-site/tunnel infection rate (reported as episodes per patient-year) in patients receiving chlorhexidine-impregnated disk

SECONDARY OUTCOMES:
Time to the first episode of exit-site/tunnel infection | one year
  days from peritoneal dialysis initiation to the time develops first exit-site/tunnel infection
peritonitis rate | one year
  Peritonitis rate (reported as episodes per patient-year) in patients receiving chlorhexidine-impregnated disk
time to first episode of peritonitis | one year
  days from peritoneal dialysis initiation to the time develops first episode of peritonitis
Peritoneal dialysis infection-related hospitalization | one year
  Hospitalization due to peritoneal dialysis-related infection
technique failure rate | one year
  technique failure is defined as transfer to hemodialysis for >= 30 days
adverse events | one year
  any local or systemic adverse events
mortality | one year
  all-cause mortality
patient satisfaction with the use of chlorhexidine-impregnated sponge dressing | third month of study
  Questionnaires related to the treatment with chlorhexidine-impregnated disk
comparison of the above outcomes with historical cohort using topical antibiotics cream | one year
  comparison of exit-site/tunnel infection rate, peritonitis rate, time to first episode of exit-site/tunnel infection or peritonitis, technique failure rate, hospitalization rate, adverse events, mortality with historical cohort patients using topical gentamicin cream

CONTACTS AND LOCATIONS:
Overall Officials: Htay Htay, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Htay H, Choo JCJ, Johnson DW, Pascoe EM, Jayaballa M, Oei EL, Ng LC, Wu SY, Foo MWY. Chlorhexidine-impregnated sponge dressing for prevention of catheter exit-site infection in peritoneal dialysis patients: a pilot study. Int Urol Nephrol. 2021 Apr;53(4):803-812. doi: 10.1007/s11255-020-02674-w. Epub 2020 Oct 6. PMID 33025409

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-04): https://cdn.clinicaltrials.gov/large-docs/20/NCT03406520/Prot_SAP_000.pdf